CLINICAL TRIAL: NCT00548418
Title: Phase II Trial of Topotecan, Cisplatin and Bevacizumab for Recurrent/Persistent Cervical Cancer
Brief Title: Topotecan, Cisplatin and Bevacizumab for Recurrent/Persistent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: GlaxoSmithKline (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-1098 / 201110266; GSK 107278
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Topotecan; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Cisplatin 50 mg/m2 IV day 1 of a 21 day cycle
  Topotecan 0.75 mg/m2 IV Days 1, 2, 3 of a 21 day cycle
  Bevacizumab 15 mg/kg day 1 of a 21 day cycle
  Interventions: Drug: Topotecan; Drug: Cisplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Topotecan
  Other Names: Hycamtin
Drug: Cisplatin
  Other Names: CDDP; Platin
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine whether the combination of topotecan, cisplatin and bevacizumab is effective in the treatment of recurrent or persistent cervical cancer

DETAILED DESCRIPTION:
Cervical cancer remains a major cause of morbidity and mortality in women. Chemoradiation has led to improvements in survival, but the prognosis for patients with recurrent, metastatic cervical cancer remains poor. There is the need for more effective treatments for the management of recurrent/persistent cervical cancer. Angiogenesis appears to play an important role in cervical cancer development and progression, therefore VEGF inhibition appears to be a rationale therapeutic strategy for cervical cancer. There is increasing evidence that combining an anti-angiogenic agent with either cytotoxic chemotherapy or radiation enhances anti-tumor activity. This study combines the current most active chemotheraputic regimen for cervical cancer (cisplatin + topotecan) with an anti-angiogenic agent.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or persistent squamous, adenosquamous or adenocarcinoma of the uterine cervix not amenable to curative treatment with surgery and/or radiotherapy
* No prior therapy (radiation, chemotherapy, hormonal therapy or immunotherapy) for recurrence or persistence. May have received platinum in combination with radiation as part of up-front treatment or adjuvant treatment
* Must have measurable disease as defined by RECIST criteria
* Must have at least one "target lesion" to assess response
* Performance status of 0 or 1
* Patients with ureteral obstruction must undergo stent or nephrostomy tube placement prior to study entry
* At least 4 weeks must have elapsed since prior treatment
* Age >= 18 years
* Patients of childbearing potential must have a negative pregnancy test, use effective means of contraception
* Signed informed consent
* Bone marrow function: ANC >= 1500/ul; platelets >= 100,000 /ul
* Renal function: creatinine <= 1,5 X ULN (if > 1.5 creatinine clearance must be > 60 ml/min)
* Hepatic function: bilirubin <= 1.5 X ULN, AST and alkaline phosphatase <= 2.5 X ULN
* Neurologic function: neuropathy < CTC grade 1
* Coagulation: PT INR <= 1.5

Exclusion Criteria:

* Evidence of sepsis or severe infection
* Prior therapy for recurrence
* Patients with serious, non-healing wound, ulcer or bone fracture
* Patients with history or evidence of nervous system disease, including primary brain tumor, brain metastases, seizure not controlled with standard medical therapy, CVA, stroke, TIA or subarachnoid hemorrhage within 6 months of 1st date of treatment on study
* Patients with history of other invasive malignancy (treatment within last 5 years) other than non-melanoma skin cancer
* Patient with clinically significant cardiovascular disease defined as:
* Inadequately controlled hypertension (systolic > 150 and/or diastolic > 100 on antihypertensive medications); prior history of hypertensive crisis or hypertensive encephalopathy
* Unstable angina within 6 months of enrollment
* NYHA Grade II or greater congestive heart failure
* Serious cardiac arrythmia requiring medication
* Grade 2 or greater peripheral vascular disease; claudication within 6 months
* History of myocardial infarction within 6 months
* Previously diagnosed coagulopathy, disseminated intravascular coagulopathy, immune thrombocytopenia purpura, thrombotic thrombocytopenia purpura or tumor involving major vessels
* Significant vascular disease: aortic aneurysm, aortic dissection
* Active thromboembolic disease: pulmonary embolism, deep venous thrombosis
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to day 1 of study; anticipation of need for major surgical procedure during course of the study
* Minor surgical procedure other than central venous access placement, within 7 days prior to day 1 of study
* Patients with proteinuria - patients with urine protein of 1+ on dipstick or >=30 mg/dl at baseline should undergo UPCR; patients with UPCR of >=1.0 should be excluded
* Patients who are pregnant or lactating
* No prior investigational agent within 30 days or planned participation in an experimental drug study
* Patients whose circumstances do not permit completion of study or required follow-up
* Prior therapy with bevacizumab or topotecan. Prior platinum therapy allowed as part of initial treatment
* History of abdominal fistula, GI perforation or intra-abdominal abscess within 6 months prior to study enrollment.
* Known hypersensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Mutch, M.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - Duke Cancer Institute, Durham, North Carolina
  - The Ohio State University College of Medicine, Columbus, Ohio

REFERENCES:
- [Derived] Zighelboim I, Wright JD, Gao F, Case AS, Massad LS, Mutch DG, Powell MA, Thaker PH, Eisenhauer EL, Cohn DE, Valea FA, Alvarez Secord A, Lippmann LT, Dehdashti F, Rader JS. Multicenter phase II trial of topotecan, cisplatin and bevacizumab for recurrent or persistent cervical cancer. Gynecol Oncol. 2013 Jul;130(1):64-8. doi: 10.1016/j.ygyno.2013.04.009. Epub 2013 Apr 13. PMID 23591400
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment to the study opened to participants on 02/20/07 and enrollment to the study was closed to participants on 11/07/11.
Groups:
- Treatment (Cisplatin, Topotecan, Bevacizumab): Cisplatin 50 mg/m2 IV day 1 of a 21 day cycle
  Topotecan 0.75 mg/m2 IV Days 1, 2, 3 of a 21 day cycle
  Bevacizumab 15 mg/kg day 1 of a 21 day cycle
Period: Overall Study
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
Performance status [Number; unit: participants] — GOG/Zubrod Description
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activitiy but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work
  2. = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. = Completely disabled
  participants
    0 | 14
    1 | 13
Disease stage [Number; unit: participants] — Stage I: The cancer has grown into the cervix, but it is not growing outside the uterus. The cancer has not spread to nearby lymph nodes or distant sites.
  Stage II: The cancer has grown beyond the cervix and uterus, but hasn't spread to the walls of the pelvis or the lower part of the vagina.
  Stage III: The cancer has spread to the lower part of the vagina or the walls of the pelvis. The cancer may be blocking the ureters. It has not spread to nearby lymph nodes or distant sites.
  Stage IV:The cancer has spread to nearby organs or other parts of the body.
  participants
    I | 9
    II | 8
    III | 8
    IV | 2
Histologic type [Number; unit: participants]
  Squamous cell | 18
  Adenocarcinoma | 9
Grade [Number; unit: participants] — 1. well differentiated
  2. moderately differentiated
  3. poorly differentiated
  participants
    1 | 2
    2 | 11
    3 | 14
Prior hysterectomy [Number; unit: participants]
  No | 22
  Yes | 5

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Activity as Measured by Surviving Progression-free
Description: Defined as the period from study entry until documentation of disease progression, death, or date of last contact, whichever occurred first.
Time Frame: Progression-free survival at 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Number analyzed (Participants) | 27
percentage of participants | 59

2. Secondary Outcome: Overall Survival
Description: Defined as time from study entry until death from any cause or date of last contaqct.
Time Frame: Until death (follow-up ranged from 1.7 months to 33.4 months)
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Number analyzed (Participants) | 27
months | 13.2 [NA to NA] — An 80% confidence interval was calculated and ranged from 8 to 15.4.

3. Secondary Outcome: Frequency of Response as Measured by RECIST Criteria (Imaging)
Description: RECIST criteria:
  Complete response is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart.
  Partial Response is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  Progression is defined as ANY of the following - 20% increase in the sum of LD target lesions, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease, progression of existing non-target lesions
  Stable disease is any condition not meeting the above criteria
Time Frame: Tumor response measured prior to every other cycle of therapy (range of follow-up to measure overall response was 1.6-9.5 months)
Population: 26 participants were evaluable for response.
Measure: Number; unit: participants
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Number analyzed (Participants) | 26
participants
  Complete response | 1
  Partial response | 8
  Stable disease | 10
  Progressive disease | 7

4. Secondary Outcome: Correlate Patterns of Gene Expression as Assessed by Microarrays
Time Frame: Correlative studies when specimens available
Population: None of the correlative studies were performed as the investigator and institution which originally offered to do those assays actually did not participate in accrual to this study. We also did not collect specimens on all patients entered on study.
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlate Hypoxia Inducible Factor 1 (HIF-1) and Hypoxia Induced Gene Expression as Measured by Laboratory Studies
Time Frame: When specimens available
Population: as for outcome 4
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment through 30 days following the end of treatment.
Arm/Group | Treatment (Cisplatin, Topotecan, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 12/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cisplatin, Topotecan, Bevacizumab) (N=27)
Esophageal stenosis (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Elevated creatinine (Investigations) | 1
Blood clot/DVT (Vascular disorders) | 2
Small bowel obstruction (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Infection - catheter (Infections and infestations) | 1
Bladder spasm (Renal and urinary disorders) | 1
Bone fracture (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Sudden cardiovascular collapse (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cisplatin, Topotecan, Bevacizumab) (N=27)
Leukopenia (Investigations) | 25
Neutropenia (Investigations) | 21
Thrombocytopenia (Investigations) | 26
Anemia (Blood and lymphatic system disorders) | 27
Allergy (Immune system disorders) | 3
Auditory (Ear and labyrinth disorders) | 1
Cardiovascular (Cardiac disorders) | 15
Coagulation (Investigations) | 9
Constitutional (Investigations) | 26
Dermatologic (Skin and subcutaneous tissue disorders) | 14
Endocrine (Endocrine disorders) | 1
Gastrointestinal (Gastrointestinal disorders) | 26
Genitourinary/renal (Renal and urinary disorders) | 13
Hemorrhage (Vascular disorders) | 6
Infection (Infections and infestations) | 12
Lymphatic (Blood and lymphatic system disorders) | 7
Metabolic (Metabolism and nutrition disorders) | 26
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3
Neurologic (Nervous system disorders) | 15
Visual (Eye disorders) | 1
Pain (General disorders) | 24
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes